CLINICAL TRIAL: NCT04352764
Title: Use of the ANTIBODY BASED LATERAL FLOW IMMUNOASSAY TESTS FOR SARSCoV-2 THAT CAUSES CORONAVIRUS DISEASE 2019 (COVID-19) - Evaluation of Patients and Healthcare Providers in the Confines of Healthcare Settings
Brief Title: ANTIBODY BASED TESTS FOR SARSCoV-2 COVID-19) - Evaluation of Patients and Healthcare Providers in the Confines of Healthcare Settings
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: TCAI_COVID-19
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CoronaCideTM COVID-19 IgM/IgG Rapid Test and Premier Biotech COVID-19 IgM/IgG Rapid Test — The tests are being distributed under section IV.D of the current United States Food and Drug Administration (FDA) policies for diagnostic tests for coronavirus disease 2019. The test is available under an emergency access mechanism called an Emergency Use Authorization (EUA). The EUA is supported by the Secretary of Health and Human Service's (HHS's) declaration that circumstances exist to justify the emergency use of in vitro diagnostics (IVDs) for the detection and/or diagnosis of the virus that causes COVID-19

SUMMARY:
This study will be conducted as a registry to identify asymptomatic or symptomatic persons to determine whether they carry SARS-CoV-2 antibodies.

DETAILED DESCRIPTION:
This study will be conducted as a registry to identify asymptomatic or symptomatic persons to determine whether they carry SARS-CoV-2 antibodies. The blood test data will be collected as allowed by the EUA using the CoronaCideTM COVID-19 IgM/IgG Rapid Test and the Premier Biotech COVID-19 IgM/IgG Rapid Test. Both COVID-19 IgM/IgG Rapid Tests are intended for Over-The-Counter/Professional use as a screening aid in the diagnosis of primary and secondary SARSCoV-2 infections, and are only for use under the FDA's EUA.

The RNA test data will be collected via a nasopharyngeal swab and processed using the Abbott ID NOW COVID-19 diagnostic test.

ELIGIBILITY:
Inclusion Criteria:

* Patient is Under the care of Texas Cardiac Arrhythmia, and Presenting to the hospital OR Presenting to a clinic conducted by Texas Cardiac Arrhythmia Or

  * An employee of Texas Cardiac Arrhythmia Or
  * An employee or healthcare professional working with patients receiving cardiac electrophysiology care at a hospital. Or A professional first responder to include Emergency Medical Services (EMS), Police or Fire departments.

Exclusion Criteria:

* Any person who refuses to undergo study procedures

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient under care of TCA or employee of TCA or employee or healthcare professional working with patients receiving cardiac electrophysiology care at a hospital
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-03-27 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
prevalence of COVID-19 exposure | Mar-Dec 2020
  To evaluate the prevalence of COVID-19 exposure to healthcare staff, community 1st responders and patients. and patient population within a subspecialty

SECONDARY OUTCOMES:
correlation between the test results with the presence or lack of COVID-19 symptoms or illness | Mar-Dec 2020
  correlation between the test results with the presence or lack of COVID-19 symptoms or illness
correlate pre-existing risk factors with test results and baseline symptoms | Mar-Dec 2020
  correlate pre-existing risk factors with test results and baseline symptoms
correlate subsequent healthcare utilization with test results and baseline symptoms | Mar-Dec 2020
  correlate subsequent healthcare utilization with test results and baseline symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- St. David's Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
No plans decided yet

REFERENCES:
- [Derived] Mohanty S, Lakkireddy D, Trivedi C, MacDonald B, Quintero Mayedo A, Della Rocca DG, Atkins D, Park P, Shah A, Gopinathannair R, Al-Ahmad A, Burkhardt JD, Gallinghouse GJ, Bassiouny M, Di Biase L, Kessler D, Tschopp D, Coffeen P, Horton R, Canby R, Natale A. Creating a safe workplace by universal testing of SARS-CoV-2 infection in asymptomatic patients and healthcare workers in the electrophysiology units: a multi-center experience. J Interv Card Electrophysiol. 2021 Oct;62(1):171-176. doi: 10.1007/s10840-020-00886-9. Epub 2020 Oct 1. PMID 33006086